CLINICAL TRIAL: NCT02952664
Title: Pressure Ulcer Monitoring Platform (PUMP): A Device to Monitor Patient Positioning
Brief Title: Pressure Ulcer Monitoring Platform (PUMP)
Acronym: PUMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, J. Peter Rubin, MD, Endowed Professor and Chair of Plastic Surgery, Professor of Bioengineering, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UPittsburghCCA
Record Dates: First submitted 2016-10-26; First posted 2016-11-02 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PUMP Monitoring (Experimental): A video camera will be placed in each subject room for recording the repositioning events to correlate the monitor signals with the actual subject repositioning captured by the video.
  Interventions: Behavioral: PUMP Monitoring

INTERVENTIONS:
Behavioral: PUMP Monitoring — A video camera will be placed in each subject room for recording the repositioning events to correlate the monitor signals with the actual subject repositioning captured by the video.

SUMMARY:
This study will employ two monitoring device prototypes. The devices are sensors containing accelerometers and gyroscope. The raw output data will be analyzed to determine when patients are moved or are repositioned in their beds. The data is captured within a modem which will correlate these movements with video recordings for interpretation by the research team. One sensor is wearable on the patient gown or sleepwear, and the other is placed underneath the frame of the hospital bed. The investigators propose a non-blinded trial with n=10 where all subjects will undergo the two devices. A video camera will be placed in each subject room for recording the repositioning events to correlate the monitor signals with the actual subject repositioning captured by the video. The goal of the trial is to validate the ability of each of the sensor prototypes to accurately detect when subjects are turned, in order to reduce stationary positioning which contributes to the incidence of pressure ulcers and to improve compliance with patient repositioning trials.

DETAILED DESCRIPTION:
The investigators propose a non-blinded trial with n=10 where all subjects will undergo the two devices. A video camera will be placed in each subject room for recording the repositioning events to correlate the monitor signals with the actual subject repositioning captured by the video. The goal of the trial is to validate the ability of each of the sensor prototypes to accurately detect when subjects are turned, in order to reduce stationary positioning which contributes to the incidence of pressure ulcers and to improve compliance with patient repositioning trials. The repositioning events recorded by the sensor devices will be automatically uploaded and abstracted by the research team, along with the events captured by the simultaneous video recording of patient repositioning.

ELIGIBILITY:
Inclusion Criteria:

* Subject is over 18 years of age
* Subject is immobile and/or unable to independently re-position self

Exclusion Criteria:

* Subject is under the age of 18 years
* Subject is able to independently re-position self

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Comparison of sensor output with video-recorded data | 10 hours of monitoring
  The dependent variables evaluated in this study are the measured outcomes as recorded by the devices and the signals collected from the accelerometer and gyroscope within said devices; the independent variable to be evaluated in this study is patient movement.

CONTACTS AND LOCATIONS:
Overall Officials: Patsy Simon, RN,BS,CCRC, Study Director — University of Pittsburgh; Joseph P Rubin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Mercy, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided